CLINICAL TRIAL: NCT04092608
Title: Impact of Goal-directed Versus Restrictive Fluid Therapy on Urethral Tissue Perfusion in Hepatobiliary Surgery: A Prospective Randomized Controlled Trial
Brief Title: Restrictive vs Goal Directed Fluid Therapy During Hepatobiliary Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Erasme University Hospital (Other)
Collaborators: Bicetre Hospital (Other)
Responsible Party: Principal Investigator, Alexandre Joosten, MD PhD, Principal Investigator, Erasme University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: B406201940521
Record Dates: First submitted 2019-09-12; First posted 2019-09-17 (Actual); Last update posted 2020-08-11 (Actual); Status verified 2020-08

CONDITIONS: Liver Surgery

STUDY DESIGN:
Intervention Model Description: Single center randomized controlled superiority study
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Low CVP group (restrictive group) (Active Comparator): Standard practice: the goal is to keep the CVP < 7 mmHg during surgery.
  Baseline of crystalloid of 2ml/kg/h max in all patients.
  EV 1000 monitoring device (Edwards Lifesciences, Irvine, USA) will be used but values will be blinded to the anesthesiologist in charge of the patient.
  Mean Arterial pressure (MAP) should be kept over 65mmHg during surgery (standard practice) with continuous norepinephrine infusion
  Additionnal fluid administration is given to the patient at the end of the surgery (standard practice)
  UPi is blinded in all groups
  Interventions: Procedure: LOW CVP (restrictive group)
- GDFT group (Experimental): The goal is to keep stroke volume variation below 13% during surgery with mini fluid challenge of 100 ml of balanced crystalloid using the monitoring device (Edwards Lifesciences, Irvine, USA). Of course, the values will not be blinded to the anesthesiologist in charge of the patient.
  All patients have a baseline crystalloid: 2ml/kg/h and mini fluid challenges per 100 ml as described above.
  Mean Arterial pressure (MAP) should be kept over 65mmHg during surgery (standard practice) with continuous norepinephrine infusion
  UPi is blinded in all groups
  Interventions: Procedure: GDFT

INTERVENTIONS:
Procedure: GDFT — The titration of fluid will be based on stroke volume variation. The goal is to maintain this variable < 13% during surgery with multiple mini fluid challenge of 100 ml of balanced crystalloid.
  Arms: GDFT group
Procedure: LOW CVP (restrictive group) — Goal = CVP < 7mmHg and only 2 ml/kg/h max during surgery.
  Arms: Low CVP group (restrictive group)

SUMMARY:
"Restrictive" fluid management is usually the current standard practice for patients undergoing liver surgery. The general idea is to maintain a low central venous pressure in order to decrease blood loss and improve the quality of the surgical field. However, this strategy , considered as rather "restrictive", can be associated with patient's harm, mainly acute kidney injury.

Today, Goal directed fluid therapy (GDFT) is a well accepted strategy to optimize fluid administration in patients undergoing major surgery which aimed to maintain normovolemia without being too liberal.

The goal of this randomized controlled trial is to compare these two strategies on Urethral Perfusion index measured with a new IKORUS UP probe (Foley catheter made smarter with embedded photoplethysmographic sensing technology).

DETAILED DESCRIPTION:
Restrictive fluid administration aiming at maintaining a low central venous pressure (low-CVP) during liver surgery has always been considered as a "gold standard" strategy because it decrease blood loss and improve the quality of the surgical field. However, this strategy , rather "restrictive", can be associated with patient harm (mainly AKI).

Today, Goal directed fluid therapy (GDFT) is a well accepted strategy to optimize fluid administration in patients undergoing major surgery.Some studies have shown that this strategy is feasible for such patient population.

There is currently a lack of data supporting the advantage of one strategy over the other in this patient population.While a restrictive fluid strategy can advantage the surgeon, it can also disadvantage the patient as in order to avoid hypotension, vasopressors administration is required. If the patient is hypovolemic, such strategy may cause acute kidney injury.

The goal of this randomized controlled trial is to compare these two strategies on Urethral Perfusion index measured with a new Foley catheter with embedded photoplethysmographic sensing technology). This new technology allows for continuous and easy monitoring of urethral tissue perfusion

The investigators hypothesis is that patients in the GDFT group will have better Urethral Perfusion index (uPI) during surgery (via a better cardiac blood flow optimization) compared to patients in the restrictive (low CVP) group.

ELIGIBILITY:
Inclusion Criteria:

-All adults patients undergoing a liver surgery and equipped with a cardiac output monitoring device

Exclusion Criteria:

-Atrial fibrillation

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-09-04 (Actual); Primary Completion 2020-07-30 (Actual); Study Completion 2020-07-30 (Actual)

PRIMARY OUTCOMES:
Urethral Perfusion index | during surgery
  average of the Urethral Perfusion index values

SECONDARY OUTCOMES:
Urethral Perfusion index | during surgery
  average of the Urethral Perfusion index values during the first 15-30 minutes of the surgery
Urethral Perfusion index | during surgery
  average of the Urethral Perfusion index values during the last 15-30 minutes of the surgery
Amount of fluid during surgery | during surgery
  amount of crystalloid received during the surgery
Amount of vasopressors | during surgery
  amount of vasopressors received during surgery
Stroke volume index | during surgery
  average of stroke volume index during surgery
stroke volume variation | during surgery
  average of stroke volume variation during surgery
cardiac index | during surgery
  average of cardiac index during surgery
incidence of acute kidney injury | At postoperative day 7
  incidence of acute kidney injury measured with the KDIGO classification
length of stay in the hospital | Postoperative day 30
  length of stay in the hospital
Incidence of postoperative complications | Postoperative day 30
  Incidence of postoperative complications

CONTACTS AND LOCATIONS:
Overall Officials: Alexandre Joosten, MD PhD, Principal Investigator — ERASME
Locations (1):
- Erasme Hospital, Brussels, Brussel-hoofdstad, Belgium

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chirnoaga D, Coeckelenbergh S, Ickx B, Van Obbergh L, Lucidi V, Desebbe O, Carrier FM, Michard F, Vincent JL, Duranteau J, Van der Linden P, Joosten A. Impact of conventional vs. goal-directed fluid therapy on urethral tissue perfusion in patients undergoing liver surgery: A pilot randomised controlled trial. Eur J Anaesthesiol. 2022 Apr 1;39(4):324-332. doi: 10.1097/EJA.0000000000001615. PMID 34669645